CLINICAL TRIAL: NCT03512496
Title: Examining the Metabolic and Genetic Impacts of Acute Energy Drink Consumption in Youth
Brief Title: Metabolic and Genetic Impacts of Energy Drinks in Youth
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: REB14-1093
Record Dates: First submitted 2018-04-05; First posted 2018-04-30 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2018-04

CONDITIONS: Nutrition; Pediatric Obesity; Pediatric; Caffeine; Metabolism Disorder, Glucose; Health Behavior; Glucose Intolerance
Keywords: Energy Drink; Pediatric; Metabolism; Glucose; Caffeine; Obesity; Nutrition; Metabolomics; Health Behavior; Glucose Intolerance
MeSH Terms: conditions — Pediatric Obesity; Glucose Metabolism Disorders; Health Behavior; Glucose Intolerance; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, crossover design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomized, double blind, crossover design

ARMS (3):
- Acute energy drink - Control (Placebo Comparator): Coloured Water was given 40 min prior to the OGTT test.
  Interventions: Dietary Supplement: Acute energy drink - Placebo
- Acute energy drink - Caffeine (Active Comparator): Sugar Free energy drink at 5mg/kg caffeine was given 40 min prior to OGTT test.
  Interventions: Dietary Supplement: Acute energy drink - Caffein
- Acute energy drink- Decaf (Sham Comparator): Sugar free decaf energy drink (vitamins only) was given 40 min prior to OGTT test. Amount of drink was same as that of Caffeine
  Interventions: Dietary Supplement: Acute energy drink - Decaf

INTERVENTIONS:
Dietary Supplement: Acute energy drink - Placebo — Colored water
  Arms: Acute energy drink - Control
Dietary Supplement: Acute energy drink - Caffein — Sugar free energy drink at 5mg/kg caffeine
  Arms: Acute energy drink - Caffeine
Dietary Supplement: Acute energy drink - Decaf — Sugar free decaf energy drink (vitamins only)
  Arms: Acute energy drink- Decaf

SUMMARY:
Caffeine containing energy drinks (CCED) are beverages that typically contain mixtures of simple sugars, caffeine and may contain vitamin, mineral and/or herbal preparations. In Canada, the consumption of CCEDs among adolescents is a regular occurrence and a common part of the everyday diet. Contributing to the obesity epidemic in youth is the consumption of energy drinks; yet no data on the metabolic responses to CCEDs exists. This study will examine the metabolic implications of CCED consumption in adolescents, aged 13-19 years. The investigators hypothesize that CCEDs will impair glucose tolerance by ~30% in lean adolescents and the primary cause of the insulin resistance will be caffeine. Obese individuals will experience a similar level of glucose impairment, but a greater rise in blood glucose compared to their lean counterparts (i.e. higher starting glucose level). For many, this additional, caffeine-induced rise will expose them to hyperglycemia, putting some individuals in the glucose intolerant or transient diabetic range. It is hypothesized that continued metabolic insult resulting from CCEDs may predispose susceptible individuals to chronic metabolic diseases later in life. The investigators will also examine the genetic basis of caffeine-induced glucose intolerance. This gene-diet interaction could explain why caffeine may be much more metabolically harmful for some individuals compared to others. The study of 'metabolomics' will also be utilized to analyze caffeine and caffeine metabolites such as theobromine, theophylline, and xanthine. This will be accomplished using Nuclear Magnetic Resonance (NMR) spectroscopy. Results from this study will have the potential to alter current perceptions that CCED are 'harmless' and will have far reaching implications for both medical professionals and legislators alike.

DETAILED DESCRIPTION:
This study will recruit male and female adolescents (aged 13-19y). Eligible participants will be booked for an initial visit where parental consent (where necessary ie. under 18 years of age) will be obtained; individuals will then be screened for overall health status. Self-report questionnaires will be administered to participants and will include information on stage of physical development (Tanner Staging), medical history, ethnicity, caffeine use (including CCEDs), gaming, physical activity and smoking status (iPad based). In the second, third and fourth visits, subjects will arrive following a 24-48h abstention from caffeine, alcohol and vigorous exercise and an overnight fast (8h). Participants will undergo three modified oral glucose tolerance tests (OGTT), following administration of either a water placebo (control), a caffeine-free CCED (control) or a caffeine containing CCED (5mg/kg caffeine) in a randomly assigned, double-blind, crossover design. Briefly, subjects will arrive and a baseline blood sample will be obtained (numbing cream will be offered). This will be immediately followed by administration of the treatment. Following a 30min absorption period, a standard OGTT (75g Trutol) will be administered. Additional blood samples will be obtained at 0, 30, 45, 60, 90, and 120min and assessed for glucose, insulin, fatty acids and C-peptide employing standard chemistry procedures. A peripheral IV will be used to obtain the 7 samples reducing needle pokes to one, ideally. Trials will be separated by at least 1wk, but not more than 4wk. Blood samples collected during the OGTT (all time points) will be assessed for metabolic and satiety signally hormone responses (ie. insulin). All subjects will also be asked to provide a saliva sample for genetic analysis. Genetic analysis will be performed by the company 23 & Me. Subjects will also be asked to provide a midstream urine sample 30 minutes prior to the completion of the OGTT (90min time point +/10 mins). This is to allow for the analysis of caffeine and caffeine metabolites present in the urine, which will give insight into how caffeine is metabolized and excreted differently among individuals.

ELIGIBILITY:
Inclusion Criteria:

* Male and female: Current data indicates no hormonal (menstrual cycle) or sex influence on caffeine pharmacokinetics or caffeine-induced insulin resistance.
* Aged 13-19: This age group has been shown to be key consumers of caffeinated energy drinks, and this study is specifically looking at the effects of these beverages in those of adolescent age.
* Lean and Obese: Individuals will be listed as obese if their Body Mass Index is greater or equal to the 85th percentile.

Exclusion Criteria:

* Participants will be excluded if they have underlying medical conditions affecting glucose tolerance, for example, inhaled steroid use, pancreatitis, diabetes, glucose intolerance etc. Any underlying condition affecting glucose tolerance would negatively skew results.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-01 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance | 120 min
  Participants will undergo an oral glucose tolerance test(OGTT), following administration of either a water placebo(control), a caffeine-free CCED or a caffeine-containing CCED.

SECONDARY OUTCOMES:
Metabolomics | 120 min
  Metabolomics will be assessed in serum collected at all time points of OGTT to analyze metabolic responses.

OTHER OUTCOMES:
Incretins | 120 min
  Incretin responses in terms of Area under the Curve (AUC) will be analyzed.
Genetic interactions | 120 min
  Genetic interactions to responses using comprehensive genotyping for polymorphism at defined loci.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada